CLINICAL TRIAL: NCT04597242
Title: Expanded Access Study of a Single Dose of Exebacase in Addition to Antistaphylococcal Antibiotics for the Treatment of Persistent Methicillin-Resistant Staphylococcus Aureus (MRSA) Bloodstream Infections (Including Right Sided Endocarditis) in Patients Who Are Hospitalized With Coronavirus Disease 2019 (COVID-19)
Brief Title: Expanded Access Study of Exebacase in COVID-19 Patients With Persistent MRSA Bacteremia
Status: No longer available | Type: Expanded Access
Sponsor: ContraFect (Industry)
Responsible Party: Sponsor
Other Study IDs: CF-301-107
Record Dates: First submitted 2020-10-20; First posted 2020-10-22 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2021-09

CONDITIONS: MRSA Bloodstream Infection; MRSA Bacteremia; MRSA Right-sided Endocarditis; Covid19
MeSH Terms: conditions — COVID-19 | interventions — exebacase

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Exebacase — Patients will receive a single IV infusion of exebacase in addition to antistaphylococcal antibiotics prescribed by the treating physician. Patients with normal renal function or mild renal impairment will be administered a dose of 18 mg of exebacase; patients with moderate or severe renal impairment will be administered a dose of 12 mg; patients with end-stage renal disease, including those on hemodialysis, will be administered a dose of 8 mg.

SUMMARY:
This is an open-label, expanded access study of exebacase used in addition to antistaphylococcal antibiotics in adult patients with persistent methicillin-resistant Staphylococcus aureus (MRSA) bloodstream infections (BSI), including right-sided endocarditis (R-IE), who are hospitalized with coronavirus disease 2019 (COVID-19). Patients with left-sided endocarditis (L-IE) are excluded. Patients will receive a single dose of exebacase. Patients will continue to receive antistaphylococcal antibiotics as prescribed by the treating physician. Exebacase Phase 3 study sites (Study CF-301-105) may participate in this Expanded Access study (Study CF-301-107).

Exebacase, a direct lytic agent, is an entirely new treatment modality against S. aureus. Exebacase is a recombinantly-produced, purified cell wall hydrolase enzyme that results in rapid bacteriolysis, potent biofilm eradication, synergy with antibiotics, low propensity for resistance, and the potential to suppress antibiotic resistance when used together with antibiotics. Exebacase represents a first-in-field, first-in-class treatment with the potential to improve clinical outcome when used in addition to standard-of-care antibiotics to treat S. aureus BSI including IE.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older.
* Hospitalized with known COVID-19 infection confirmed by positive diagnostic test.
* Not eligible for the exebacase Phase 3 study (CF-301-105).
* Blood cultures positive for MRSA for ≥3 days.
* Patient is not pregnant or breastfeeding and is not of reproductive potential or agrees to remain abstinent or use contraception if of reproductive potential.

Exclusion Criteria:

* Known or suspected left-sided IE.
* Intubated for COVID-19.
* Presence of prosthetic valve or cardiac valve support ring, or presence of known infected orthopedic hardware, prosthetic joint, or cardiac device.
* Known or suspected brain abscess or meningitis.
* Participation in an investigational study or expanded access protocol for another antistaphylococcal antibacterial agent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - CF-301-107 Study Site, Butte, Montana
  - Cf 301-107, Toledo, Ohio